CLINICAL TRIAL: NCT02459132
Title: A Phase II Randomized Trial of High-Intensity Aerobic Interval Training and Surrogate Markers of Cardiovascular Disease in a Population-based Sample of Testicular Cancer Survivors
Brief Title: High-Intensity Aerobic Interval Training in Testicular Cancer Survivors
Acronym: HIITTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HREBA.CC-14-0183
Record Dates: First submitted 2015-05-21; First posted 2015-06-01 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2016-09

CONDITIONS: Cardiovascular Diseases; Testicular Neoplasms
Keywords: High-intensity interval training; VO2peak; Brachial flow-mediated dilation; Carotid-femoral pulse wave velocity; Carotid intima-media thickness; Carotid distensibility; Respiratory sinus arrhythmia
MeSH Terms: conditions — Cardiovascular Diseases; Testicular Neoplasms; Arrhythmia, Sinus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Group (Experimental): Subjects in the exercise group will attend supervised exercise sessions three times a week, for 12 weeks. The exercise intervention will consist of uphill walking or jogging on a treadmill between 50% and 95% of VO2peak for 35 minutes (including a 5-minute warm up and cool down). The participants will complete four, 4-minute, high-intensity intervals at 85-95% of VO2peak. The work period intervals will be interspersed with three, 3-minute periods of active recovery at an intensity below that of their ventilatory threshold.
  Interventions: Behavioral: High-intensity aerobic interval exercise
- Usual Care (No Intervention): The usual care group will not receive an intervention, and they will be asked to maintain baseline physical activity levels throughout the observation period.

INTERVENTIONS:
Behavioral: High-intensity aerobic interval exercise — See arm/group description
  Arms: Exercise Group

SUMMARY:
This study evaluates the impact of a supervised 12-week high-intensity aerobic interval exercise program (versus a self-directed exercise usual care group) on traditional and novel cardiovascular disease risk factors and surrogate markers of cardiovascular- and overall-mortality in a population-based sample of testicular cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed history of testicular cancer

Exclusion Criteria:

* Not sufficiently ambulatory to complete the first two stages of the aerobic exercise test.
* Have a psychiatric condition which impairs their ability to perform the required volume and intensity of exercise.
* Have any uncontrolled cardiovascular condition (i.e. heart disease, hypertension, diabetes, arrhythmia).
* Report performing any weekly vigorous intensity aerobic exercise in the past month.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-07; Primary Completion 2016-09 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Peak aerobic capacity (relative VO2peak) | Baseline and within 7 days of completing the 12-week intervention
  ml O2/kg/min

SECONDARY OUTCOMES:
Peak aerobic capacity (absolute VO2peak) | Baseline and within 7 days of completing the 12-week intervention
  L/min
Postexercise 1-minute heart rate recovery | Baseline and within 7 days of completing the 12-week intervention
  change in beats/min
Heart rate | Baseline and within 7 days of completing the 12-week intervention
  beats/min
Systolic blood pressure | Baseline and within 7 days of completing the 12-week intervention
  mmHg
Diastolic blood pressure | Baseline and within 7 days of completing the 12-week intervention
  mmHg
Respiratory sinus arrhythmia | Baseline and within 7 days of completing the 12-week intervention
  beats/min
Average carotid intima-media thickness | Baseline and within 7 days of completing the 12-week intervention
  mm
Maximal carotid intima-media thickness | Baseline and within 7 days of completing the 12-week intervention
  mm
Carotid distensibility | Baseline and within 7 days of completing the 12-week intervention
  10-3/kPa
Carotid diameter | Baseline and within 7 days of completing the 12-week intervention
  mm
Brachial flow-mediated dilation | Baseline and within 7 days of completing the 12-week intervention
  percent dilation
Brachial diameter | Baseline and within 7 days of completing the 12-week intervention
  mm
Velocity time integral | Baseline and within 7 days of completing the 12-week intervention
  cm
Shear stress during reactive hyperemia | Baseline and within 7 days of completing the 12-week intervention
  dynes/cm2
Carotid-femoral pulse wave velocity | Baseline and within 7 days of completing the 12-week intervention
  m/s
Femoral-toe pulse wave velocity | Baseline and within 7 days of completing the 12-week intervention
  m/s
Fibrinogen | Baseline and within 7 days of completing the 12-week intervention
  g/L
High-sensitivity C-reactive protein | Baseline and within 7 days of completing the 12-week intervention
  mg/L
Total cholesterol | Baseline and within 7 days of completing the 12-week intervention
  mmol/L
High-density lipoprotein | Baseline and within 7 days of completing the 12-week intervention
  mmol/L
Low-density lipoprotein | Baseline and within 7 days of completing the 12-week intervention
  mmol/L
Total cholesterol : high-density lipoprotein ratio | Baseline and within 7 days of completing the 12-week intervention
  ratio
Triglycerides | Baseline and within 7 days of completing the 12-week intervention
  mmol/L
Fasting glucose | Baseline and within 7 days of completing the 12-week intervention
  mmol/L
Testosterone | Baseline and within 7 days of completing the 12-week intervention
  nmol/L
Framingham Risk Score | Baseline and within 7 days of completing the 12-week intervention
  10 year CVD risk %
Vascular age | Baseline and within 7 days of completing the 12-week intervention
  years
Modifiable CVD Risk Factor Score | Baseline and within 7 days of completing the 12-week intervention
  Number (max 24)

OTHER OUTCOMES:
Health-related quality of life | Baseline, within 7 days of completing the 12-week intervention, and approximately 3 months after the post-intervention testing
  Short form 36
Depression | Baseline, within 7 days of completing the 12-week intervention, and approximately 3 months after the post-intervention testing
  Centre for epidemiologic studies depression scale
Fatigue | Baseline, within 7 days of completing the 12-week intervention, and approximately 3 months after the post-intervention testing
  Functional Assessment of Cancer Therapy - Fatigue
Sleep Quality | Baseline, within 7 days of completing the 12-week intervention, and approximately 3 months after the post-intervention testing
  Global Pittsburg Sleep Quality Index
Anxiety | Baseline, within 7 days of completing the 12-week intervention, and approximately 3 months after the post-intervention testing
  Spielberger State Anxiety Scale
Stress | Baseline, within 7 days of completing the 12-week intervention, and approximately 3 months after the post-intervention testing
  Perceived Stress Scale
Self-Esteem | Baseline, within 7 days of completing the 12-week intervention, and approximately 3 months after the post-intervention testing
  Rosenberg Self-Esteem Scale

CONTACTS AND LOCATIONS:
Overall Officials: Kerry S Courneya, PhD, Principal Investigator — University of Alberta

REFERENCES:
- [Derived] Adams SC, DeLorey DS, Davenport MH, Stickland MK, Fairey AS, North S, Szczotka A, Courneya KS. Effects of high-intensity aerobic interval training on cardiovascular disease risk in testicular cancer survivors: A phase 2 randomized controlled trial. Cancer. 2017 Oct 15;123(20):4057-4065. doi: 10.1002/cncr.30859. Epub 2017 Jul 14. PMID 28708930